CLINICAL TRIAL: NCT02937129
Title: Clinical Accuracy and Reliability of Infrared Tympanic Thermometer in an Adult Emergency Department
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Fangge Deng, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 20151A010093
Record Dates: First submitted 2016-10-10; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Fever
Keywords: Infrared tympanic thermometer; Axillary thermometer; Mercury glass thermometer; Adult emergency department
MeSH Terms: conditions — Fever; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of this study was to determine the accuracy of an infrared thermometer compared to the gold standard, mercury-in-glass thermometer. The secondary aim was to compare tympanic and axillary temperature measurements by evaluating agreement and correlation to determine whether an infrared tympanic thermometer can replace an axillary mercury thermometer in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Above 37.5°C measured by axillary mercury thermometer

Exclusion Criteria:

1. otitis external/media
2. soft-tissue infection over the axillary fossa and forehead
3. complete occlusion by earwax
4. severe illness
5. trauma

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Febrile patients defined by a cut off of 37.5°C measured by axillary mercury thermometer were enrolled. Patients who meet the exclusion criteria were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The body temperatures of fever patients measured by the infrared tympanic thermometer | up to 5 months
  1. Fever patients were measured by the infrared tympanic thermometer in the emergency department.
  2. Their tympanic temperatures were obtained from both sides of the body three times.
  3. Use statistical methods to evaluate the relevance and consistency between the tympanic temperatures and gold standard temperatures(measured by the glass mercury thermometer).